CLINICAL TRIAL: NCT03456726
Title: A Phase 2 Study of Tazemetostat in Relapsed or Refractory B-cell Non-Hodgkin's Lymphoma With EZH2 Gene Mutation
Brief Title: Study of Tazemetostat in Participants With Relapsed or Refractory B-cell Non-Hodgkin's Lymphoma With EZH2 Gene Mutation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E7438-J081-206
Record Dates: First submitted 2018-03-06; First posted 2018-03-07 (Actual); Results first posted 2022-12-16 (Actual); Last update posted 2022-12-16 (Actual); Status verified 2021-04

CONDITIONS: Relapsed or Refractory B-cell Non-Hodgkin's Lymphoma
Keywords: EZH2 gene mutation; Tazemetostat; Diffuse large B-cell lymphoma; Follicular lymphoma
MeSH Terms: conditions — Recurrence; Lymphoma, B-Cell; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular | interventions — tazemetostat

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- FL with EZH2 gene mutation (Experimental): Participants with follicular lymphoma (FL) with the EZH2 gene mutation will receive oral tazemetostat at a starting dose of 800 milligrams (mg) twice daily (1600 mg total daily dose) by continuous regimen, no less than 8 hours between doses.
  Interventions: Drug: Tazemetostat
- DLBCL with EZH2 gene mutation (Experimental): Participants with diffuse large B-cell lymphoma (DLBCL) with the EZH2 gene mutation will receive oral tazemetostat at a starting dose of 800 mg twice daily (1600 mg total daily dose) by continuous regimen, no less than 8 hours between doses.
  Interventions: Drug: Tazemetostat

INTERVENTIONS:
Drug: Tazemetostat — Tazemetostat will be provided as a 200 mg oral tablet.

SUMMARY:
This is a multicenter, open-label, Phase 2 study to assess the efficacy and safety of tazemetostat in participants with relapsed or refractory B-cell non-Hodgkin's lymphoma (NHL) with EZH2 gene mutation.

ELIGIBILITY:
Inclusion Criteria:

* Participants with histological diagnosis of B-cell non-Hodgkin's lymphoma (NHL) as follows:

  * Cohort 1: Follicular lymphoma (FL)
  * Cohort 2: Diffuse large B-cell lymphoma (including primary mediastinal B-cell lymphoma and transformed FL)
* Participants who have confirmed EZH2 gene mutation of tumor in central laboratory
* Participants who have measurable disease
* Participants who had previous therapy with systemic chemotherapy and/or antibody therapy and for which no standard therapy exists
* Participants who had progressive disease or did not have response (complete response or partial response) in previous systemic therapy, or relapsed or progressed after previous systemic therapy
* Participants with Eastern Cooperative Oncology Group performance status of 0 to 1
* Participants with life expectancy of ≥3 months from starting study drug administration
* Participants with adequate renal, liver, and bone marrow function
* Male and female participants ≥20 years of age at the time of informed consent
* Participants who has provided written consent to participate in the study

Exclusion Criteria:

* Participants with prior exposure to EZH2 inhibitor
* Participants with a history or a presence of central nerves invasion
* Participants with malignant pleural effusion, cardiac effusion, or ascites retention
* Participants with allogeneic stem cell transplantation
* Participants with medical need for the continued use of potent inhibitors of Cytochrome P450 3A (CYP3A)or potent inducer of CYP3A (including St. John's wort)
* Participants with significant cardiovascular impairment

  · Participants with prolongation of corrected QT interval using Fridericia's formula to > 480 milliseconds (msec)
* Participants with venous thrombosis or pulmonary embolism within the last 3 months before starting study drug
* Participants with complications of hepatic cirrhosis, interstitial pneumonia or pulmonary fibrosis
* Participants with active infection requiring systemic therapy
* Women of childbearing potential or man of impregnate potential who don't agree that both the participant and his/her partner will use a medically effective method for contraception for periods from before informed consent to during the clinical study and 30 days later (for males 90 days later) from last administration of study drug
* Woman who are pregnant or breastfeeding
* Participants who were deemed as inappropriate to participate in the study by the investigator or sub-investigator
* Have any prior history of T-cell lymphoblastic lymphoma/T-cell acute lymphoblastic leukemia or myeloid malignancies, including myelodysplastic syndrome

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-04-09 (Actual); Primary Completion 2021-12-17 (Actual); Study Completion 2021-12-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (28):
- Japan (28):
  - 1004 Eisai Trial Site, Nagoya, Aichi-ken
  - 1029 Eisai Trial Site, Nagoya, Aichi-ken
  - 1020 Eisai Trial Site, Ōta, Gunma
  - 1007 Eisai Trial Site, Sapporo, Hokkaido
  - 1019 Eisai Trial Site, Kobe, Hyōgo
  - 1005 Eisai Trial Site, Tsukuba, Ibaraki
  - 1002 Eisai Trial Site, Isehara, Kanagawa
  - 1028 Eisai Trial Site, Yokohama, Kanagawa
  - 1021 Eisai Trial Site, Sendai, Miyagi
  - 1013 Eisai Trial Site, Sayama, Osaka
  - 1006 Eisai Trial Site, Suita, Osaka
  - 1027 Eisai Trial Site, Suntou-gun, Shizuoka
  - 1026 Eisai Trial Site, Bunkyo-ku, Tokyo
  - 1001 Eisai Trial Site, Chuo-ku, Tokyo
  - 1025 Eisai Trial Site, Koto-ku, Tokyo
  - 1017 Eisai Trial Site, Minato-ku, Tokyo
  - 1022 Eisai Trial Site, Aomori
  - 1010 Eisai Trial Site, Chiba
  - 1012 Eisai Trial Site, Fukuoka
  - 1016 Eisai Trial Site, Fukuoka
  - 1011 Eisai Trial Site, Hiroshima
  - 1024 Eisai Trial Site, Kumamoto
  - 1003 Eisai Trial Site, Kyoto
  - 1008 Eisai Trial Site, Kyoto
  - 1023 Eisai Trial Site, Nagasaki
  - 1009 Eisai Trial Site, Okayama
  - 1015 Eisai Trial Site, Osaka
  - 1018 Eisai Trial Site, Yamagata

REFERENCES:
- [Derived] Izutsu K, Ando K, Nishikori M, Shibayama H, Goto H, Kuroda J, Kato K, Imaizumi Y, Nosaka K, Sakai R, Abe M, Hojo S, Nakanishi T, Rai S. Tazemetostat for relapsed/refractory B-cell non-Hodgkin lymphoma with EZH2 mutation in Japan: 3-year follow-up for a phase II study. Int J Hematol. 2024 Nov;120(5):621-630. doi: 10.1007/s12185-024-03834-9. Epub 2024 Aug 23. PMID 39179948

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 28 investigative sites in Japan from 09 April 2018 to 17 December 2021.
Pre-assignment Details: A total of 100 participants were screened, of which 80 were screen failures and only 20 participants were eligible to enter the study and received the study treatment.
Groups:
- Participants With Follicular Lymphoma: Participants with follicular lymphoma (FL) with the enhancer of zeste homolog 2 (EZH2) gene mutation received oral tazemetostat tablet at a starting dose of 800 milligrams (mg) twice daily (1600 mg total daily dose) in Cycle 1 and 2 and subsequent cycles (Cycle length=28 days) by continuous regimen, no less than 8 hours between doses until disease progression (PD), development of unacceptable toxicity, participant's requests to discontinue, withdrawal of consent, or study termination by the sponsor.
- Participants With Diffuse Large B-cell Lymphoma: Participants with diffuse large B-cell lymphoma (DLBCL) with the EZH2 gene mutation received oral tazemetostat at a starting dose of 800 mg twice daily (1600 mg total daily dose) in Cycle 1 and 2 and subsequent cycles (Cycle length=28 days) by continuous regimen, no less than 8 hours between doses until PD, development of unacceptable toxicity, participant's requests to discontinue, withdrawal of consent, or study termination by the sponsor.
Period: Overall Study
Arm/Group | Participants With Follicular Lymphoma | Participants With Diffuse Large B-cell Lymphoma
Started | 17 | 3
Completed | 0 | 0
Not Completed | 17 | 3
Not completed — Disease Progression | 6 | 1
Not completed — Adverse Event | 4 | 2
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Discontinued from study due to switch to commercial tazemetostat | 6 | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set included participants who received at least 1 administration of the study drug.
Groups:
- Participants With Follicular Lymphoma: Participants with FL with the EZH2 gene mutation received oral tazemetostat tablet at a starting dose of 800 mg twice daily (1600 mg total daily dose) in Cycle 1 and 2 and subsequent cycles (Cycle length=28 days) by continuous regimen, no less than 8 hours between doses until PD, development of unacceptable toxicity, participant's requests to discontinue, withdrawal of consent, or study termination by the sponsor.
- Participants With Diffuse Large B-cell Lymphoma: Participants with DLBCL with the EZH2 gene mutation received oral tazemetostat at a starting dose of 800 mg twice daily (1600 mg total daily dose) in Cycle 1 and 2 and subsequent cycles (Cycle length=28 days) by continuous regimen, no less than 8 hours between doses until PD, development of unacceptable toxicity, participant's requests to discontinue, withdrawal of consent, or study termination by the sponsor.
- Total: Total of all reporting groups
Arm/Group | Participants With Follicular Lymphoma | Participants With Diffuse Large B-cell Lymphoma | Total
Number analyzed (Participants) | 17 | 3 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.8 (9.28) | 74.7 (7.23) | 67.1 (9.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 2 | 11
  Male | 8 | 1 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 17 | 3 | 20
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 17 | 3 | 20
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) Based on Independent Reviewer Assessment
Description: ORR was defined as percentage of participants with confirmed best overall response (BOR) of complete response (CR) or partial response (PR) using independent reviewer assessment based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. BOR of CR and PR was confirmed by a subsequent CR assessment and CR or PR assessment. CR: disappearance of all measurable, non-measurable lesions and no unequivocal new lesions. Any pathological lymph nodes (target or non-target) had to be reduced in short axis to less than (<) 10 millimeter (mm). PR: at least a 30 percent (%) decrease in sum of diameters (SOD) of target lesions, taking as reference the baseline SOD and there are no unequivocal new lesions, and no progression of non-target disease. The 2-sided 95% confidence interval (CI) was calculated by Clopper-Pearson method.
Time Frame: From date of first dose of study drug administration to date of PD or death, whichever occurred first (up to 3 years 4 months)
Population: The efficacy analysis set included efficacy evaluable participants who received at least 1 administration of the study drug and who has appropriate tumor assessment data of Screening 2 (Screening 2 was conducted in this study to confirm the other eligibility for study treatment) and post-baseline.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Participants With Follicular Lymphoma | Participants With Diffuse Large B-cell Lymphoma
Number analyzed (Participants) | 17 | 3
percentage of participants | 76.5 [50.1 to 93.2] | 100.0 [29.2 to 100.0]

2. Primary Outcome: ORR Based on Investigator Assessment
Description: ORR was defined as percentage of participants with confirmed BOR of CR or PR using investigator assessment based on RECIST 1.1. BOR of CR and PR was confirmed by a subsequent CR assessment and CR or PR assessment. CR: disappearance of all measurable, non-measurable lesions and no unequivocal new lesions. Any pathological lymph nodes (target or non-target) had to be reduced in short axis <10 mm. PR: at least a 30% decrease in SOD of target lesions, taking as reference the baseline SOD and there are no unequivocal new lesions, and no progression of non-target disease. The 2-sided 95% CI was calculated by Clopper-Pearson method.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Participants With Follicular Lymphoma | Participants With Diffuse Large B-cell Lymphoma
Number analyzed (Participants) | 17 | 3
percentage of participants | 70.6 [44.0 to 89.7] | 66.7 [9.4 to 99.2]

3. Secondary Outcome: Progression-free Survival (PFS) Based on Independent Reviewer Assessment
Description: PFS was assessed by independent reviewer assessment based on RECIST 1.1. PFS was defined as the time from the date of the first dose of study drug to the date of the first documentation of PD or death, whichever occurred first. PD for target lesion, a minimum 20% increase and a minimum 5 mm absolute increase in SOD compared to nadir, or PD for non-target lesion(s) or unequivocal new lesion(s). Nadir: Lowest measure SOD of target lesion at any time point from baseline onward. The 95% CI was calculated using Kaplan-Meier estimate.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Participants With Follicular Lymphoma | Participants With Diffuse Large B-cell Lymphoma
Number analyzed (Participants) | 17 | 3
months | NA [12.9 to NA] — Median and upper limit of 95% CI was not estimable due to insufficient PFS events observed. | 15.7 [5.3 to NA] — The upper limit of 95% CI was not estimable due to insufficient PFS events observed.

4. Secondary Outcome: PFS Based on Investigator Assessment
Description: PFS was assessed by investigator assessment based on RECIST 1.1. PFS was defined as the time from the date of the first dose of study drug to the date of the first documentation of PD or death, whichever occurred first. PD for target lesion, a minimum 20% increase and a minimum 5 mm absolute increase in SOD compared to nadir, or PD for non-target lesion(s) or unequivocal new lesion(s). Nadir: Lowest measure SOD of target lesion at any time point from baseline onward. The 95% CI was calculated using Kaplan-Meier estimate.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Participants With Follicular Lymphoma | Participants With Diffuse Large B-cell Lymphoma
Number analyzed (Participants) | 17 | 3
months | NA [18.4 to NA] — Median and upper limit of 95% CI was not estimable due to insufficient PFS events observed. | 26.7 [5.3 to NA] — The upper limit of 95% CI was not estimable due to insufficient PFS events observed.

5. Secondary Outcome: Duration of Response (DOR) Based on Independent Reviewer Assessment
Description: DOR: time from date of confirmation of the first response and the date of confirmation of the PD using independent reviewer assessment as per RECIST 1.1. BOR of CR and PR was confirmed by subsequent CR assessment and CR or PR assessment, respectively at least 4 weeks later. CR: disappearance of all measurable, non-measurable lesions and no unequivocal new lesions. Any pathological lymph nodes had to be reduced in short axis to <10 mm. PR: at least 30% decrease in SOD of target lesions, taking as reference the baseline SOD, there are no unequivocal new lesions, and no progression of non-target disease. PD for target lesion, a minimum 20% increase and a minimum 5mm absolute increase in SOD compared to nadir, or PD for non-target lesions or unequivocal new lesions. Nadir: Lowest measure SOD of target lesions at any time point from baseline onward. The 95% CI was calculated using Kaplan-Meier estimate.
Time Frame: From the date of first confirmed objective response (OR) to PD or death due to confirmed PR or CR (up to 3 years 4 months)
Population: The efficacy analysis set included efficacy evaluable participants who received at least 1 administration of the study drug and who has appropriate tumor assessment data of Screening 2 (Screening 2 was conducted in this study to confirm the other eligibility for study treatment) and post-baseline. Here, Overall number of participants analyzed signifies participants who had OR (CR or PR) as per Independent Reviewer Assessment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Participants With Follicular Lymphoma | Participants With Diffuse Large B-cell Lymphoma
Number analyzed (Participants) | 13 | 3
months | NA [11.0 to NA] — Median and upper limit of 95% CI was not estimable due to insufficient number of responders with events observed. | 13.8 [1.6 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of responders with events observed.

6. Secondary Outcome: DOR Based on Investigator Assessment
Description: as for outcome 5
Time Frame: From the date of first confirmed OR to PD or death due to any cause for those participants with a confirmed PR or CR (up to 3 years 4 months)
Population: The efficacy analysis set included efficacy evaluable participants who received at least 1 administration of the study drug and who has appropriate tumor assessment data of Screening 2 (Screening 2 was conducted in this study to confirm the other eligibility for study treatment) and post-baseline. Here, Overall number of participants analyzed signifies participants who had OR (CR or PR) as per Investigator Assessment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Participants With Follicular Lymphoma | Participants With Diffuse Large B-cell Lymphoma
Number analyzed (Participants) | 12 | 2
months | 35.8 [22.1 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of responders with events observed. | NA [21.1 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of responders with events observed.

7. Secondary Outcome: Time to Response (TTR) Based on Independent Reviewer Assessment
Description: TTR was defined as the time from the first dose of the study drug to date of first observation of CR or PR using independent reviewer assessment based on RECIST 1.1. CR: disappearance of all measurable, non-measurable lesions and no unequivocal new lesions. Any pathological lymph nodes (target or non-target) had to be reduced in short axis to <10 mm. PR: at least a 30% decrease in SOD of target lesions, taking as reference the baseline SOD and there are no unequivocal new lesions, and no progression of non-target disease.
Time Frame: From the date of first dose until date of first observation of CR or PR (up to 3 years 4 months)
Population: as for outcome 5
Measure: Median (Full Range); unit: months
Arm/Group | Participants With Follicular Lymphoma | Participants With Diffuse Large B-cell Lymphoma
Number analyzed (Participants) | 13 | 3
months | 3.64 [1.8 to 10.1] | 3.70 [1.9 to 7.4]

8. Secondary Outcome: TTR Based on Investigator Assessment
Description: TTR was defined as the time from the first dose of the study drug to date of first observation of CR or PR using investigator assessment based on RECIST 1.1. CR: disappearance of all measurable, non-measurable lesions and no unequivocal new lesions. Any pathological lymph nodes (target or non-target) had to be reduced in short axis to <10 mm. PR: at least a 30% decrease in SOD of target lesions, taking as reference the baseline SOD and there are no unequivocal new lesions, and no progression of non-target disease.
Time Frame: From the date of first dose until date of first observation of CR or PR (up to 3 years 4 months)
Population: as for outcome 6
Measure: Median (Full Range); unit: months
Arm/Group | Participants With Follicular Lymphoma | Participants With Diffuse Large B-cell Lymphoma
Number analyzed (Participants) | 12 | 2
months | 4.59 [1.8 to 7.5] | 5.56 [5.5 to 5.6]

9. Secondary Outcome: Number of Participants With Any Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: TEAE is defined as an AE that emerged during time from the first dose of study drug to 30 days after the participant's last dose. An AE was any untoward medical occurrence in participant administered with an investigational product. An SAE was any untoward medical occurrence that at any dose: resulted in death; life threatening; requires participant hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity; was a congenital anomaly/birth defect (in the child of a participant who was exposed to the study drug).
Time Frame: From the first dose of study drug to 30 days after the last dose (up to 3 years 5 months)
Population: The safety analysis set included participants who received at least 1 administration of the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Follicular Lymphoma | Participants With Diffuse Large B-cell Lymphoma
Number analyzed (Participants) | 17 | 3
Participants
  TEAEs | 17 | 3
  SAEs | 8 | 1

ADVERSE EVENTS:
Time Frame: From the first dose of study drug to 30 days after the last dose (up to 3 years 5 months)
Arm/Group | Participants With Follicular Lymphoma | Participants With Diffuse Large B-cell Lymphoma
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/3
Serious Adverse Events (participants affected / at risk) | 8/17 | 1/3
Other Adverse Events (participants affected / at risk) | 17/17 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants With Follicular Lymphoma (N=17) | Participants With Diffuse Large B-cell Lymphoma (N=3)
Mechanical ileus (Gastrointestinal disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Atypical pneumonia (Infections and infestations) | 1 | 0
Periodontitis (Infections and infestations) | 1 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants With Follicular Lymphoma (N=17) | Participants With Diffuse Large B-cell Lymphoma (N=3)
Lymphopenia (Blood and lymphatic system disorders) | 5 | 0
Neutropenia (Blood and lymphatic system disorders) | 3 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 0
Anaemia (Blood and lymphatic system disorders) | 2 | 0
Hypochromic anaemia (Blood and lymphatic system disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Conjunctival haemorrhage (Eye disorders) | 1 | 1
Cataract (Eye disorders) | 1 | 0
Visual impairment (Eye disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 5 | 0
Stomatitis (Gastrointestinal disorders) | 5 | 0
Nausea (Gastrointestinal disorders) | 3 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Epigastric discomfort (Gastrointestinal disorders) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0
Large intestine polyp (Gastrointestinal disorders) | 1 | 0
Tooth disorder (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 1 | 1
Malaise (General disorders) | 2 | 0
Non-cardiac chest pain (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Hypogammaglobulinaemia (Immune system disorders) | 1 | 0
Nasopharyngitis (Infections and infestations) | 7 | 1
Upper respiratory tract infection (Infections and infestations) | 5 | 0
Herpes simplex (Infections and infestations) | 2 | 0
Influenza (Infections and infestations) | 2 | 0
Pneumonia (Infections and infestations) | 2 | 0
Urinary tract infection (Infections and infestations) | 2 | 0
Bronchitis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Impetigo (Infections and infestations) | 1 | 0
Oral herpes (Infections and infestations) | 1 | 0
Paronychia (Infections and infestations) | 1 | 0
Periodontitis (Infections and infestations) | 1 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Postoperative delirium (Injury, poisoning and procedural complications) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 0
Traumatic fracture (Injury, poisoning and procedural complications) | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 5 | 0
Blood creatinine increased (Investigations) | 3 | 0
Weight decreased (Investigations) | 3 | 0
Amylase increased (Investigations) | 2 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood pressure decreased (Investigations) | 1 | 0
Blood zinc decreased (Investigations) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0
Immature granulocyte count increased (Investigations) | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Tendon disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Dysgeusia (Nervous system disorders) | 9 | 1
Dizziness (Nervous system disorders) | 0 | 1
Muscle spasticity (Nervous system disorders) | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Visual field defect (Nervous system disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Hypertonic bladder (Renal and urinary disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 4 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 1
Eczema (Skin and subcutaneous tissue disorders) | 2 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 0
Keloid scar (Skin and subcutaneous tissue disorders) | 1 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
Phlebitis (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-01-29): https://cdn.clinicaltrials.gov/large-docs/26/NCT03456726/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-31): https://cdn.clinicaltrials.gov/large-docs/26/NCT03456726/SAP_001.pdf